CLINICAL TRIAL: NCT06655480
Title: Effect on Clinical Status, Structural and Functional Cardiac Parameters and Myocardial Fibrosis of Triple Combination Therapy With a Sodium-glucose Cotransporter 2 Inhibitor, Angiotensin Receptor/Neprilysin Inhibitor and Mineralocorticoid Receptor Antagonist in Patients With Advanced HFpEF
Brief Title: Triple Combination Therapy (ARNI, SGLT2i, MRA) in Advanced HFpEF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Collaborators: Lomonosov Moscow State University Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 124020200111-6
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: HFpEF; LVDD; Myocardial Fibrosis
Keywords: HFpEF; HF; left ventricular hypertrophy; diastolic dysfunction; cardiac reserves; LV filling pressures; myocardial fibrosis
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [ARNI + SGLTi + AMR] (Experimental): Patients will receive combination therapy with ARNI, gliflozin and AMR
  Interventions: Drug: [ARNI + SGLTi + AMR]
- [SGLTi + previously taken RAAS blocker] (Active Comparator): Patients will receive combination therapy with gliflozin and previously taken RAAS blocker
  Interventions: Drug: [SGLTi + previously taken RAAS blocker]

INTERVENTIONS:
Drug: [ARNI + SGLTi + AMR] — Empagliflozin 10mg tablet, Valsartan+Sacubitril 100-200-400 mg tablet, Finerenone 20-40 mg tablet
  Arms: [ARNI + SGLTi + AMR]
Drug: [SGLTi + previously taken RAAS blocker] — Empagliflozin 10mg tablet, previously taken RAAS inhibitor
  Arms: [SGLTi + previously taken RAAS blocker]

SUMMARY:
Patients with advanced heart failure with preserved ejection fraction (HFpEF) will be randomly assigned in open-label multicenter study to receive triple combination therapy with [angiotensin receptor/neprilysin inhibitor [ARNI] + sodium-glucose cotransporter 2 inhibitor [SGLTi] + mineralocorticoid receptor antagonist [MRA]) or with individualized medical therapy [SGLTi + renin-angiotensin system inhibitor [RASi] [angiotensin receptor blocker [ARB] or angiotensin-converting enzyme inhibitor [ACE-I]), and will be treated for 52 weeks

DETAILED DESCRIPTION:
HFpEF has a signiﬁcant morbidity and mortality, and the therapeutic options for HFpEF are limited. According to the results of clinical HFpEF trials, SGLTis and MRA can improve prognosis (EMPEROR-preserved, DELIVER, FINEARTS-HF trials); and ARNI can reduce the risk of hospitalization due to exacerbation of heart failure (PARAGON-HF trial). There is also clinical and experimental evidence of anti-inflammatory and antifibrotic effects in SGLTi, MRA and ARNI. However, there are currently no randomized clinical trials evaluating the efficacy of the combination therapy with all these drugs in HFpEF. The investigators suppose that triple combination therapy with [ARNI + SGLTi + AMR] in HFpEF will have a pronounced, rapid and safe positive clinical and haemodynamic effect primarily through its effect on fibrosis and inflammation in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and data informed consent;
2. Symptoms and signs of HF;
3. LV ejection fraction > 50%;
4. NT-proBNP > 300 pg/mL (for patients with atrial fibrillation NT-proBNP > 900 pg/mL)
5. LV diastolic dysfunction II-III grade OR

LV diastolic dysfunction I grade and at least 2 out of 4:

* Е/е' > 14
* LAVi > 34 ml/m2 (for those with persistent atrial fibrillation > 40 ml/m2)
* PASP > 35 mm Hg or TR velocity > 2.8 m/sec
* LV mass index > 95 g/m2 for women / > 115 g/m2 for men or LV interventricular septum or posterior wall thickness ≥ 1.1 sm OR

Chronic atrial fibrillation and at least 3 out of 4:

* Е/е' > 11
* E-wave velocity > 100 sm/s
* TR velocity > 2.8 sm/s
* DT ≤ 160 ms

Exclusion Criteria:

1. Evidence of myocardial ischemia during stress echocardiography;
2. Significant lesions of main coronary arteries;
3. Atrial fibrillation with resting HR > 110 beats/min;
4. Continuous (>90 days) treatment with ARNI, SGLTi and/or AMR within 12 months prior to screening. The last administration of these drugs must be at least 30 days prior to randomization. Treatment with these drugs should not be interrupted for the purpose of inclusion in the study.
5. Coronary bypass surgery, stroke or TIA within the last 3 months of screening;
6. Myocardial infarction or myocardial revascularization within the last 3 months of screening;
7. Systolic blood pressure < 90 mmHg or ≥ 180 mmHg at screening or randomization;
8. Genetic forms of HFpEF (HCM, amyloidosis, Fabry disease, glycogen storage diseases etc.);
9. Peripartum cardiomyopathy, chemotherapy-induced cardiomyopathy, viral myocarditis, isolated right-sided HF without left-sided structural disease, constrictive pericarditis, significant pericardial effusion;
10. Dyspnea due to non-cardiac causes such as pulmonary disease, anemia, severe obesity, primary valvular, or myocardial diseases;
11. Significant lung disease (severe lung disease requiring home oxygen or chronic oral steroid therapy);
12. Primary pulmonary artery hypertension;
13. Significant left sided structural valve disease;
14. Anemia (Hb < 100 g/L);
15. Obesity (body mass index > 50 kg/m2);
16. Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (CKD-EPI);
17. Impaired liver function (serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 × upper limit of normal);
18. Addison's disease;
19. Known hypersensitivity to medications used the in the study;
20. Non-cardiac conditions that complicate/exclude participation in the study;
21. Diseases associated with isolated LV insufficiency (idiopathic pulmonary hypertension, chronic thromboembolic pulmonary hypertension, etc.);
22. Serum/plasma potassium >5.0 mmol/L at screening or randomization or a history of hyperkalemia or acute renal failure during AMR treatment for >7 consecutive days leading to discontinuation of AMR treatment.
23. For patients with diabetes mellitus:

    * Type 1 diabetes mellitus;
    * Presence of more than 4 episodes of moderate hypoglycemia within the past month or at least one episode of severe hypoglycemia within the past year;
    * Glycated hemoglobin level > 9% or <6%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-18 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial extracellular volume (MRI) | 52 weeks
  Difference in myocardial extracellular volume assessed by MRI data between 52 weeks after baseline and at baseline
Change in 6-minute walking distance (6MWD) | 52 weeks
  Difference in distance walked during 6-minute walking test (6MWT) between 52 weeks after baseline and at baseline
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) | 52 weeks
  Difference in NT-proBNP plasma levels between 52 weeks after baseline and at baseline
Change in average E/e' ratio and tricuspid regurgitation velocity | 52 weeks
  Difference in E/e' ratio and tricuspid regurgitation velocity assessed by echocardiography both at rest and at peak exercise during diastolic stress test (DST) between 52 weeks after baseline and at baseline
Change in left atrial volume index (LAVi) | 52 weeks
  Difference in LAVi assessed by echocardiography between 52 weeks after baseline and at baseline

SECONDARY OUTCOMES:
Change in left ventricular mass index (LVMi) | 52 weeks
  Difference in LVMi assessed by MRI between 52 weeks after baseline and at baseline
Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) score | 52 weeks
  Difference in Minnesota Living with Heart Failure Questionnaire (MLHFQ, potential scoring range between 0 and 105; higher scores mean a worse outcome) score between 52 weeks after baseline and at baseline
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 52 weeks
  Difference in Kansas City Cardiomyopathy Questionnaire (KCCQ; a range of possible subscale scores is from 0 to 100, with 100 representing the least burden of symptoms. The total KCCQ score represents the mean of the three subscale scores) score between 52 weeks after baseline and at baseline
Change in biomarkers of inflammation and fibrosis | 52 weeks
  Difference in plasma levels of inflammatory and fibrosis biomarkers (hsCRP, GDF-15, PICP, galectin-3, MCP-1) between 52 weeks after baseline and at baseline
Change in cardiac hemodynamic reserves - LV contractile | 52 weeks
  Difference in cardiac hemodynamic reserves (LV contractile) during DST between 52 weeks after baseline and at baseline
Change in cardiac hemodynamic reserves - LV diastolic | 52 weeks
  Difference in cardiac hemodynamic reserves (LV diastolic) during DST between 52 weeks after baseline and at baseline
Change in cardiac hemodynamic reserves - LA reservoir | 52 weeks
  Difference in cardiac hemodynamic reserves (LA reservoir) during DST between 52 weeks after baseline and at baseline
Change in cardiac hemodynamic reserves - cardiac chronotropic | 52 weeks
  Difference in cardiac hemodynamic reserves (cardiac chronotropic) during DST between 52 weeks after baseline and at baseline
Change in cardiac hemodynamic reserves - RV contractile | 52 weeks
  Difference in cardiac hemodynamic reserves (RV contractile) during DST between 52 weeks after baseline and at baseline